CLINICAL TRIAL: NCT07381283
Title: Clinical and Radiographic Evaluation of Immediate Versus Delayed Loading of Dental Implants at the Anterior Maxilla
Brief Title: Immediate Versus Delayed Loading of Dental Implants in the Anterior Maxilla
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Suez Canal University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 706/2023
Record Dates: First submitted 2026-01-25; First posted 2026-02-02 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: Partial Edentulism of the Maxilla; Dental Implant Loading; Tooth Loss in the Anterior Maxilla
Keywords: Dental Implants; Immediate Loading; Delayed Loading; Maxillary Implants; Anterior Maxilla; Partial Edentulism; Implant Stability; Osseointegration
MeSH Terms: interventions — Dental Implants

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Delayed Loading Group (Active Comparator): Participants in this group received a single dental implant placed in the anterior maxilla. A total of eight implants were placed and restored using a delayed loading protocol, with prosthetic loading performed six months after implant placement.
  Interventions: Device: Dental Implant
- Immediate Loading Group (Experimental): Participants in this group received a single dental implant placed in the anterior maxilla. A total of eight implants were placed and immediately loaded with provisional restorations. After six months, the provisional restorations were replaced with definitive fixed restorations.
  Interventions: Device: Dental Implant

INTERVENTIONS:
Device: Dental Implant — Endosseous dental implants placed in the anterior maxilla and restored using either immediate or delayed loading protocols.

SUMMARY:
This interventional comparative clinical study was conducted to evaluate and compare the clinical stability and radiographic outcomes of immediate versus delayed loading of dental implants placed in the anterior region of the maxilla. Immediate loading protocols have been shown to improve oral health-related quality of life and patient satisfaction; however, their influence on implant stability and osseointegration remains an area of ongoing investigation.

A total of sixteen dental implants were placed and the participants were randomly allocated into two equal groups using a computer-generated randomization method (www.Randomizer.org). In Group I (control group), eight implants were placed and restored following a delayed loading protocol, with prosthetic loading performed six months after implant placement. In Group II (study group), eight implants were placed and immediately loaded with provisional polymethyl methacrylate (PMMA) restorations. After six months, the provisional restorations were replaced with definitive fixed prostheses.

Preoperative planning of implant placement was performed using cone beam computed tomography (CBCT). Clinical evaluation of implant stability was carried out using the Osstell device, while radiographic assessment of peri-implant bone density and marginal bone changes was performed using standardized indirect digital radiographs. Radiographic evaluations were obtained immediately after implant placement and at six months postoperatively. The clinical and radiographic outcomes of both loading protocols were compared to assess implant stability and osseointegration.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 20-55 years
* Both genders
* Healthy individuals (ASA I) without systemic diseases
* Patients with one or more missing teeth in the anterior maxilla

Exclusion Criteria:

* Pregnant or lactating women, or females with osteoporosis
* Patients with harmful oral habits such as bruxism or smoking
* Poor oral hygiene
* Gingival or periodontal diseases with severe vertical or horizontal bone loss
* Teeth with periapical or lateral infections or lesions

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2024-02-03 (Actual); Primary Completion 2025-05-21 (Actual); Study Completion 2025-10-12 (Actual)

PRIMARY OUTCOMES:
Implant Stability (ISQ) | Baseline (immediately after implant placement) and 6 months postoperatively
  Clinical stability of dental implants was assessed using the Osstell device. The implant stability quotient (ISQ) was measured immediately after implant placement and at 6 months postoperatively. ISQ scores range from 1-100, with scores ≥70 indicating high stability, 60-69 medium stability, and <60 low stability.
Peri-implant Bone Density | Baseline, 3 months, 6 months
  Bone density around the implants was measured using standardized direct paralleling digital periapical radiographs and analyzed with IDRISI Kilimanjaro software. Two zones were evaluated: the osseointegration zone near the implant border and the surrounding bone interface. Measurements were recorded immediately postoperatively and at 3 and 6 months.

SECONDARY OUTCOMES:
Postoperative Pain (Visual Analog Scale, VAS) | 1, 3, and 7 days postoperatively
  Patients reported the degree of pain using a 10-cm visual analog scale (VAS), where 0 = no pain and 10 = worst possible pain. Pain was assessed at 1, 3, and 7 days postoperatively.
Visual Scale of Edema | 1, 3, and 7 days postoperatively
  Facial edema was assessed using a visual grading scale: No edema, Low-grade, Intermediate-grade, and High-grade, based on visual inspection and palpation. Edema was evaluated at 1, 3, and 7 days postoperatively.

CONTACTS AND LOCATIONS:
Overall Officials: Mohamed Said Hamed, Professor, Study Chair — Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry - Suez Canal University; Asmaa Yousri Abdallah, Assistant professor, Study Director — Assistant professor of Oral Radiology, Faculty of Dentistry; Ahmed Abd elmohsen Younis, Assistant professor, Study Director — Assistant Professor of Oral and Maxillofacial Surgery, Faculty of Dentistry - Suez Canal University
Locations (1):
- Suez Canal University, Faculty of Dentistry, Ismailia, Egypt

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kim HS, Cho HA, Kim YY, Shin H. Implant survival and patient satisfaction in completely edentulous patients with immediate placement of implants: a retrospective study. BMC Oral Health. 2018 Dec 18;18(1):219. doi: 10.1186/s12903-018-0669-1. PMID 30563482
- [Background] Gallucci GO, Hamilton A, Zhou W, Buser D, Chen S. Implant placement and loading protocols in partially edentulous patients: A systematic review. Clin Oral Implants Res. 2018 Oct;29 Suppl 16:106-134. doi: 10.1111/clr.13276. PMID 30328194
- [Background] Fischer K, Stenberg T, Hedin M, Sennerby L. Five-year results from a randomized, controlled trial on early and delayed loading of implants supporting full-arch prosthesis in the edentulous maxilla. Clin Oral Implants Res. 2008 May;19(5):433-41. doi: 10.1111/j.1600-0501.2007.01510.x. Epub 2008 Mar 26. PMID 18371094
- [Background] Eliasziw M, Young SL, Woodbury MG, Fryday-Field K. Statistical methodology for the concurrent assessment of interrater and intrarater reliability: using goniometric measurements as an example. Phys Ther. 1994 Aug;74(8):777-88. doi: 10.1093/ptj/74.8.777. PMID 8047565
- [Background] Cohen, J. 1988. Statistical power analysis for the behavioral sciences. Hillsdale, New Jersey: Lawrence Erlbaum Associates.
- [Background] Bergkvist G, Sahlholm S, Nilner K, Lindh C. Implant-supported fixed prostheses in the edentulous maxilla. A 2-year clinical and radiological follow-up of treatment with non-submerged ITI implants. Clin Oral Implants Res. 2004 Jun;15(3):351-9. doi: 10.1111/j.1600-0501.2004.01017.x. PMID 15142099
- [Background] Bergkvist G, Nilner K, Sahlholm S, Karlsson U, Lindh C. Immediate loading of implants in the edentulous maxilla: use of an interim fixed prosthesis followed by a permanent fixed prosthesis: a 32-month prospective radiological and clinical study. Clin Implant Dent Relat Res. 2009 Mar;11(1):1-10. doi: 10.1111/j.1708-8208.2008.00094.x. Epub 2008 Apr 1. PMID 18384401